CLINICAL TRIAL: NCT05883215
Title: Effects of Social Media Usage on Pain Catastrophizing and Disease Impact in Female Patients With Fibromyalgia Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Collaborators: Başakşehir Çam & Sakura City Hospital (Other Government); Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: FMS1
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female Patients Diagnosed with Fibromyalgia Syndrome: Female patients who give consent to participate and are diagnosed with fibromyalgia syndrome.
  Interventions: Other: Pain catastrophizing scale; Other: Beck Anxiety Inventory; Other: Social Media Use Integration Scale; Other: Fibromyalgia Impact Questionnaire

INTERVENTIONS:
Other: Pain catastrophizing scale — The pain catastrophizing scale is a self-report questionnaire used to assess an individual's tendency to engage in catastrophic thinking when experiencing pain. It measures the extent to which a person magnifies, feels helpless, and feels unable to cope with pain. The scale typically consists of several items that ask individuals to rate the degree to which they experience specific thoughts or emotions related to pain catastrophizing, such as "I worry all the time about whether the pain will end" or "I feel like I can't stand it anymore." Participants provide responses on a Likert scale indicating the intensity or frequency of their agreement with each statement. The scale helps researchers and healthcare professionals gain insights into an individual's cognitive and emotional responses to pain, which can have implications for pain management strategies and overall well-being.
Other: Beck Anxiety Inventory — Beck Anxiety Inventory" (BAI), which is designed to measure the severity of anxiety symptoms in individuals. The BAI is a self-report questionnaire consisting of 21 items that assess various symptoms of anxiety, such as nervousness, fear, and physiological manifestations of anxiety. Participants rate the intensity of their symptoms over the past week on a scale ranging from 0 (not at all) to 3 (severely). The scores obtained on the BAI can help clinicians and researchers evaluate the presence and severity of anxiety symptoms, monitor changes over time, and guide treatment decisions. It is important to note that the BAI is not a diagnostic tool but rather a measure of self-reported anxiety symptoms.
Other: Social Media Use Integration Scale — The Social Media Use Integration Scale (SMUIS) is a self-report measure that assesses the degree to which individuals integrate social media into their daily lives. It aims to capture the extent to which individuals incorporate social media use into various aspects of their routines, behaviors, and identity. The scale typically consists of items that assess factors such as the frequency and duration of social media use, the importance and impact of social media on personal relationships, the integration of social media into daily activities, and the emotional connection to social media.
Other: Fibromyalgia Impact Questionnaire — The Fibromyalgia Impact Questionnaire (FIQ) is a widely used self-report measure specifically designed to assess the impact of fibromyalgia on various aspects of a person's life. It is a multidimensional questionnaire that evaluates the physical functioning, social functioning, and overall well-being of individuals with fibromyalgia.
  The FIQ typically consists of items that ask individuals to rate the impact of fibromyalgia on their ability to perform daily activities, such as work, household chores, and recreational activities. It also assesses the severity of fibromyalgia symptoms, including pain, fatigue, sleep disturbances, and cognitive difficulties. Additionally, the questionnaire may include items related to emotional well-being, social support, and overall quality of life.

SUMMARY:
The aim of this study is to investigate the effects of social media usage on pain catastrophizing and disease impact in female individuals diagnosed with fibromyalgia syndrome.

DETAILED DESCRIPTION:
In this study, the total number of female patients obtained as a result of sample size calculations was 73, and the effect of social media use on pain catastrophizing and disease impact of patients diagnosed with fibromyalgia will be investigated. Social media use will be evaluated with the Social Media Use Integration Scale, disease impact with the Fibromyalgia Impact Questionnaire, anxiety levels with the Beck Anxiety Inventory, and pain catastrophizing level with the pain catastrophizing scale. At the same time, a form including demographic data of the patients will be filled. The results will be evaluated with the tests prescribed by the statistical expert, and correlation will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Giving consent.
* Being diagnosed with Fibromyalgia syndrome
* Being female

Exclusion Criteria:

* Not giving consent.
* Any disability or illness that may prevent filling out the form or communicating.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on gender identity.
Study Population: Female patients with fibromyalgia syndrome diagnosis who gave consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between social media use and pain catastrophizing | 1 day
  The possible correlation between the results obtained with the social media integration scale and the results obtained with the pain catastrophizing scale will be investigated with statistical methods.
Correlation between social media use and disease impact | 1 day
  The possible correlation between the results obtained with the social media integration scale and the results obtained with the fibromyalgia impact questionnaire will be investigated with statistical methods.
Correlation between social media use and anxiety | 1 day
  The possible correlation between the results obtained with the social media integration scale and the results obtained with the Beck Anxiety Inventory will be investigated with statistical methods.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Principal Investigator — Uskudar State Hospital

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data will be shared upon reasonable request by the corresponding author.